CLINICAL TRIAL: NCT05869201
Title: Double-blind Comparative Randomized Tolerability, Safety and Immunogenicity Trial of the Flu-M Quadro Tetravalent Inactivated Split Influenza Vaccine, Solution for Intramuscular Injection, FSUE SPbSRIVS FMBA of Russia, in Volunteers Aged 18-60 Years
Brief Title: Tolerability, Safety and Immunogenicity Trial of the Flu-M Quadro, Tetravalent Inactivated Split Influenza Vaccine
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: St. Petersburg Research Institute of Vaccines and Sera (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMK-II/III-02/20
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Influenza; Influenza, Human; Influenza Viral Infections; Vaccine Reaction; Vaccination; Infection
Keywords: Influenza; Flu; Vaccine; Vaccination; SPbSRIVS; Flu-M Tetra; Flu-M Quadro; Quadrivalent; Inactivated; Split
MeSH Terms: conditions — Influenza, Human; Infections | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Flu-M Quadro with preservative (Experimental): 150 volunteers were vaccinated with the Flu-M Quadro Inactivated Split Influenza Vaccine with a preservative
  Interventions: Biological: Influenza vaccine [inactivated]
- Flu-M Quadro without preservative (Experimental): 150 volunteers were vaccinated with the Flu-M Quadro Inactivated Split Influenza Vaccine without a preservative
  Interventions: Biological: Influenza vaccine [inactivated]
- Ultrix® Quadri (Active Comparator): 150 volunteers were vaccinated with Ultrix® Quadri Vaccine
  Interventions: Biological: Influenza vaccine [inactivated]

INTERVENTIONS:
Biological: Influenza vaccine [inactivated] — Solution for intramuscular injection, 0.5 ml (1 dose) Vaccination with a single dose vaccine
  Other Names: Flu-M Quadro (with a preservative)
  Arms: Flu-M Quadro with preservative
Biological: Influenza vaccine [inactivated] — Solution for intramuscular injection, 0.5 ml (1 dose) Vaccination with a single dose vaccine
  Other Names: Flu-M Quadro (without preservative)
  Arms: Flu-M Quadro without preservative
Biological: Influenza vaccine [inactivated] — Solution for intramuscular injection, 0.5 ml (1 dose) Vaccination with a single dose vaccine
  Other Names: Ultrix® Quadri
  Arms: Ultrix® Quadri

SUMMARY:
The goal of this clinical trial is to assess tolerability, safety and immunogenicity of the Flu-M Quadro vaccine as compared to the Ultrix® Quadri vaccine in volunteers aged between 18 and 60.

Participants were given Flu-M Quadro [inactivated split influenza vaccine] with preservative or Flu-M Quadro [inactivated split influenza vaccine] without preservative or Ultrix® Quadri vaccine.The volunteers of each group were vaccinated with a single dose vaccine.

Researchers assessed the tolerability, safety and immunogenicity of the Flu-M Quadro quadrivalent inactivated split influenza vaccine.

Researchers performed a comparative assessment of the tolerability, safety, and immunogenicity of the Flu-M Quadro quadrivalent inactivated split influenza vaccine and the Ultrix® Quadri vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men and women) aged 18-60;
* Written informed consent of the volunteers to participate in the clinical trial;
* Volunteers able to fulfill requirements of the protocol (i.e., fill out the patient's diary, come to follow-up visits);
* For fertile women - a negative result of the pregnancy test and consent to observe adequate methods of contraception (usage of contraceptives one month before vaccination and at least two months after vaccination). All females with childbearing potential must have a negative pregnancy test result during the screening period. In the course of the trial women should use barrier contraceptives with a reliability exceeding 90 %, or be sterile, or be in a postmenopausal state. Barrier contraceptives with a reliability exceeding 90 % of common use include cervical caps with spermicide, diaphragms with spermicide, condoms, intra-uterine spirals;
* For the men, are able to conceive - consent to use adequate contraception methods. In the course of the trial and during at least two months after vaccination, men and their sexual partners should use barrier contraceptives with a reliability exceeding 90 %, or be sterile. Barrier contraceptives with a reliability exceeding 90 % of common use include cervical caps with spermicide, diaphragms with spermicide, condoms, intra-uterine spirals;

Exclusion Criteria:

* History of influenza or ARVI or previous influenza vaccination during 9 moths before the trial;
* A serious post-vaccination reaction (temperature above 40 °C, hyperemia or edema more than 8 cm in diameter) or complications (collapse or shock-like condition that developed within 48 hours after vaccination; convulsions accompanied or not accompanied by a fever due to any previous vaccination);
* Allergic reactions to vaccine components or any previous vaccination;
* History of allergic reaction to chicken protein;
* History of Guillain-Barré syndrome (acute polyneuropathy);
* Previous vaccination with rabies vaccines less than 2 months before immunization or scheduled vaccination with rabies vaccines within 1 month after immunization with the trial vaccines;
* Use of any vaccines within 1 month before the vaccination, excluding vaccines according to the National Calendar of Preventive Vaccination, including for epidemic reasons;
* History of leukemia, tuberculosis, cancer, autoimmune diseases;
* Positive blood test results for HIV, syphilis, hepatitis B/C.
* Volunteers who received immunoglobulin or blood products or had a blood transfusion during the last three months before the trial;
* History of long-term use (more than 14 days) of immunosuppressants or other immunomodulatory drugs for six months before the trial;
* History of any confirmed or suspected immunosuppressive or immunodeficiency condition;
* History of chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine systems, the gastrointestinal tract, liver, kidneys, hematopoietic or immune systems, mental disease in the acute stage or in the decompensation stage (recovery less than 4 weeks before vaccination);
* History of progressive neurological pathology, convulsive syndrome; Diabetes mellitus, thyrotoxicosis or other diseases of the endocrine system;
* History of eczema;
* Treatment with glucocorticosteroids, including in small doses, as well as local use of drugs containing steroids (> 10 mg of prednisolone or its equivalent for more than 14 days during the last three months);
* According to the medical history, the volunteer was/is a patient of a tuberculosis dispensary and/or narcological dispensary and/or neuropsychiatric dispensary and/or other;
* History of acute infectious diseases (recovery less than 4 weeks before vaccination);
* Consumption of more than 10 units of alcoholic drinks per week or history of alcohol addiction, drug addiction or abuse of pharmaceutical products;
* Smoking of more than 10 cigarettes per day;
* Participation in another clinical trial during the last 3 months;
* Pregnancy or lactation;
* Serious concurrent illnesses or pathological conditions not listed above which, in the opinion of the investigator, could complicate the assessment of the results of the trial including pathological deviations from age norms and laboratory norms of blood and urine parameters, which are clinically significant in the opinion of the investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 450 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate for each virus strain (A (H1N1), A (H3N2) and B (Yamagata line and Victoria line)) The percentage of subjects who have a prevaccination titer of influenza haemagglutinin antibody titer (HA titer) ≤ 1:10 and a postvaccination HA titer | Screening (Days 0+5), Day 28

SECONDARY OUTCOMES:
Change from Baseline Geometric mean titer (GMT) ratio of antibodies for each virus strain (A (H1N1), A (H3N2) and B (Yamagata line and Victoria line)) | Screening (Days 0+5), Day 28
  Geometric mean titer (GMT) of antibodies in the blood serums of vaccinated participants in haemagglutination inhibition assay
Seroconversion factor for each virus strain (A (H1N1), A (H3N2) and B (Yamagata line and Victoria line)) Seroconversion factor is an increase in the geometric mean titers of antibodies at Day 28 vs. the baseline level, expressed in the fold rise | Screening (Days 0+5), Day 28
Seroprotection rate for each virus strain (A (H1N1), A (H3N2) and B (Yamagata line and Victoria line)) Seroprotection rate is the percentage of subjects with a generated protective HA titer (at least 1:40) vs. the baseline level | Screening (Days 0+5), Day 28
Incidence of influenza and ARVI | During 6 months after vaccination
  Incidence, severity, and duration of influenza and ARVI during 6 months after vaccination detected outside of the Protocol.
Incidence of immediate adverse events (allergic reactions) | 2 hours after vaccination
Incidence of local adverse events | 7 days after vaccination
Incidence of systemic adverse events | 7 days after vaccination
Incidence of other adverse reactions | Days 8 to 28 after vaccination
Incidence of severe adverse events | Days 1 to 28 after vaccination
Incidence of withdrawal of a volunteer from the trial due to development of an AE/SAE associated with the use of the trial products | Days 1-7, 14
Number of participants with abnormal physical examination findings | Screening (Days 0+5), Days 1-7, 14, 28
  Physical examination of volunteers included an interview, discovery of complaints and symptoms, when required, palpation, auscultation, percussion. During the interview, all complaints and symptoms that had developed since the last visit were identified and assessed. An examination and (when applicable) palpation, auscultation, percussion were performed for the following organs and systems: skin, mucosa, eyes, oral cavity and pharynx, lungs/chest, heart/cardiovascular system, abdominal organs, nervous system, lymph nodes, musculoskeletal system, thyroid gland. The palpation analysis of lymph nodes (submandibular, cervical, ulnar) included an assessment of their size, consistency, pain, mobility, adhesion between themselves and with surrounding tissues and skin
Number of participants with abnormal changes in vital signs - Blood pressure (BP) | Screening (Days 0+5), Days 1-7, 14, 28
  BP measurements include the systolic and diastolic blood pressure
Number of participants with abnormal changes in vital signs - Heart rate (HR) | Screening (Days 0+5), Days 1-7, 14, 28
  HR is measured using a phonendoscope at the apex of the heart during 1 minute
Number of participants with abnormal changes in vital signs - Respiratory rate (RR) | Screening (Days 0+5), Days 1-7, 14, 28
Number of participants with abnormal changes in vital signs - Body temperature | Screening (Days 0+5), Day 1 - before vaccination, 20 minutes and 2, 5-8 hours after vaccination; Days 2-7, 14, 28
  Body temperature was measured using mercury or digital thermometer, in the armpit for at least 5 minutes
Number of participants with clinically significant abnormalities - Complete blood count (CBC) | Screening (Days 0+5), Days 3, 14, 28
  Red blood cells, Hemoglobin, ESR, Differential Leukocyte Count (segmented and rod neutrophils, lymphocytes, monocytes, eosinophils, basophils), Platelets
Number of participants with clinically significant abnormalities - Biochemical blood test (BBT) | Screening (Days 0+5), Days 3, 14, 28
  ALT, AST, Alkaline phosphatase, Total Bilirubin, Total Protein, Urea, Glucose, C-reactive protein, Creatinine, Cholesterol
Number of participants with clinically significant abnormalities - Urinalysis | Screening (Days 0+5), Days 3, 14, 28
  pH, Relative Density/Specific Gravity, Protein, Glucose, Red Blood Cells, White Blood Cells
Number of participants with abnormal changes of total IgE | Screening (Days 0+5), Days 3, 14, 28
Number of participants with abnormal neurological examinations | Screening (Days 0+5), Days 1, 3 (When the interval between the screening visit and visit 1 is more than 3 days), 14, 28
Number of participants with abnormal electrocardiography results | Screening (Days 0+5), Day 3
  Standard 12-lead ECG

CONTACTS AND LOCATIONS:
Overall Officials: Ellina Ruzanova, Study Director — St. Petersburg Research Institute of Vaccines and Sera
Locations (5):
- Russia (5):
  - Federally Funded Healthcare Institution Primary Healthcare Unit No. 163,of Federal Medical and Biologic Agency (FFHI PHU No. 163, FMBA of Russia), Kol'tsovo, Novosibirsk Oblast
  - Bessalar Clinic. Clinical Trial Center Limited Liability Company (Bessalar Clinic. Clinical Trial Center LLC), Moscow
  - Federation (FSBEI of Higher Education "E. A. Wagner PSMU" of the of the Ministry of Health of the Russian Federation), Perm
  - Baltic Medicine Limited Liability Company (Baltic Medicine LLC), Saint Petersburg
  - Eco-Safety Scientific Research and Development Center Limited Liability Company (Eco-Safety Scientific Research and Development Center LLC), Saint Petersburg